CLINICAL TRIAL: NCT05664334
Title: A Phase 1 Randomized, Observer-blind, Placebo-controlled, Multi-center Trial to Evaluate the Safety and Immunogenicity of IVX-A12, a Respiratory Syncytial Virus and Human Metapneumovirus Bivalent Combination Virus-like Particle Protein Subunit Vaccine, in Healthy Adults, 60 to 75 Years of Age
Brief Title: Safety and Immunogenicity of IVX-A12 in Healthy Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Icosavax, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: ICVX-12-101
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Respiratory Syncytial Virus; Human Metapneumovirus; Bivalent Combination Virus-like Particle Protein Subunit Vaccine
MeSH Terms: interventions — MF59 oil emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- IVX-A12 Vaccine - Low Dosage Level (Experimental): Participants will receive IVX-A12 vaccine (bivalent combination formulation containing IVX-121 and IVX-241 virus-like particles [VLPs]), administered intramuscularly (IM) once on Day 0.
  Interventions: Biological: IVX-121; Biological: IVX-241
- IVX-A12 Vaccine + MF59® - Low Dosage Level (Experimental): Participants will receive IVX-A12 vaccine (bivalent combination formulation containing IVX-121 and IVX-241 VLPs), administered IM once on Day 0.
  Interventions: Biological: IVX-121; Biological: IVX-241; Other: MF59®
- IVX-A12 Vaccine - Medium Dosage Level (Experimental): Participants will receive IVX-A12 vaccine (bivalent combination formulation containing IVX-121 and IVX-241 VLPs), administered IM once on Day 0.
  Interventions: Biological: IVX-121; Biological: IVX-241
- IVX-A12 Vaccine + MF59® - Medium Dosage Level (Experimental): Participants will receive IVX-A12 vaccine (bivalent combination formulation containing IVX-121 and IVX-241 VLPs), administered IM once on Day 0.
  Interventions: Biological: IVX-121; Biological: IVX-241; Other: MF59®
- IVX-A12 Vaccine - High Dosage Level (Experimental): Participants will receive IVX-A12 vaccine (bivalent combination formulation containing IVX-121 and IVX-241 VLPs), administered IM once on Day 0.
  Interventions: Biological: IVX-121; Biological: IVX-241
- Placebo (Placebo Comparator): Participants will receive placebo, administered IM once on Day 0.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: IVX-121 — 75 mcg of IVX-121 without MF59®
  Arms: IVX-A12 Vaccine - Low Dosage Level
Biological: IVX-241 — 75 mcg of IVX-241 without MF59®
  Arms: IVX-A12 Vaccine - Low Dosage Level
Biological: Placebo — Diluent
  Arms: Placebo
Biological: IVX-121 — 75 mcg of IVX-121, without MF59®
  Arms: IVX-A12 Vaccine - High Dosage Level; IVX-A12 Vaccine - Medium Dosage Level
Biological: IVX-241 — 150 mcg IVX-241, without MF59®
  Arms: IVX-A12 Vaccine - Medium Dosage Level
Biological: IVX-241 — 225 mcg of IVX-241, without MF59®
  Arms: IVX-A12 Vaccine - High Dosage Level
Biological: IVX-121 — 75 mcg of IVX-121, with MF59®
  Arms: IVX-A12 Vaccine + MF59® - Low Dosage Level; IVX-A12 Vaccine + MF59® - Medium Dosage Level
Biological: IVX-241 — 75 mcg of IVX-241, with MF59®
  Arms: IVX-A12 Vaccine + MF59® - Low Dosage Level
Biological: IVX-241 — 150 mcg IVX-241, with MF59®
  Arms: IVX-A12 Vaccine + MF59® - Medium Dosage Level
Other: MF59® — MF59® as an adjuvant
  Arms: IVX-A12 Vaccine + MF59® - Low Dosage Level; IVX-A12 Vaccine + MF59® - Medium Dosage Level

SUMMARY:
The main purpose of this study is to evaluate the safety and immunogenicity of three dosage levels (low, medium, high) of the bivalent combination respiratory syncytial virus (RSV)/human metapneumovirus (hMPV) virus-like particle (VLP) candidate vaccine (IVX-A12), compared to placebo, when administered as a single-dose regimen in healthy older adults 60 to 75 years of age.

DETAILED DESCRIPTION:
The Phase 1 clinical trial of IVX-A12 is a randomized, observer-blinded, placebo-controlled, multi-center study designed to evaluate the safety and immunogenicity of multiple dosage levels of IVX-A12, with and without CSL Seqirus' proprietary adjuvant MF59®.

A total of up to 120 healthy older adults aged 60 to 75 years. Participants will be administered a single shot of IVX-A12, at one of three combination dosage levels below, or placebo. The overall duration of the study is up to 1 year (365 days).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female older adults 60 to 75 years of age at the time of first vaccination
* Participants with stable well-controlled chronic conditions such as hypertension without clinical exacerbation of their underlying disease within the previous 12 months
* Participants able to voluntarily give written informed consent and to comply with study procedures including follow-up to approximately 12 months after first dosing
* Body mass index (BMI) 17 to 35 kilogram per square meter (kg/m^2), inclusive, at screening
* Screening laboratory values must be within the laboratory reference ranges or deemed not clinically significant if within Grade 1 severity on the toxicity scale

Exclusion Criteria:

* Prior receipt of any investigational RSV or hMPV vaccine
* Prior receipt of another investigational medicinal product (study drug, biologic, or device) not authorized for use in the United States and European Union within the past year
* Laboratory-confirmed severe RSV or hMPV infection within the past year prior to enrollment
* Currently enrolled or plan to participate in another clinical study with an investigational agent (including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication) to be received during the study period
* Presence of high-risk comorbidities for severe RSV or hMPV disease (example, significant cardiopulmonary disease)
* Older adults meeting frail elderly criteria (older persons with medical, nutritional, cognitive, emotional, or activity impairments, as defined by the study site)
* Acute or chronic progressive, unstable or uncontrolled clinical conditions
* Acute illness, with or without fever at the time of planned vaccination
* History of hypersensitivity or serious adverse reactions to vaccines, such as anaphylaxis, Guillain-Barré, and angioedema, or any known allergies to any component of the IVX-121 and/or IVX-241 vaccine, or hypersensitivity to latex
* Abnormal function of the immune system resulting from clinical conditions including human immunodeficiency virus, chronic administration of systemic corticosteroids (oral/intravenous/IM at a dose equivalent of greater than (>) 20 milligrams (mg) prednisone in a period of more than 14 days), or administration of immunosuppressive chemotherapy, biologics, or radiotherapy within the past 3 months before study randomization
* Refusal to maintain contraceptive practices during the study, and (for women of childbearing potential) to be screened for pregnancy at specified times during the study
* Receipt of licensed inactivated vaccines including influenza vaccine within 14 days prior to study vaccine administration on Study Day 0, or with live virus vaccines within 30 days of Day 0

  1. Receipt of licensed vaccines is permitted after completion of the study Day 28 visit.
  2. Receipt of licensed COVID-19 vaccines is permitted if dosing regimen completed within 21 days prior to study vaccine administration on Day 0 or after completion of the Day 28 visit.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants With Solicited Local Reactions and Systemic AEs | Within 7 days After the Dose (From Day 0 to Day 6)
Proportion of Participants With Unsolicited AEs | Up to 28 days After the Dose (From Day 0 to Day 28)
Proportion of Participants With RSV/A, RSV/B, hMPV/A and hMPV/B Neutralizing Antibodies (NAb) | At Day 28
Proportion of Participants With RSV and hMPV Immunoglobulin G (IgG) Prefusion F Protein-specific Antibody Titers | At Day 28
  RSV and hMPV IgG prefusion F protein-specific antibody titers as measured by enzyme-linked immunosorbent assays (ELISAs).

SECONDARY OUTCOMES:
Proportion of Participants With at Least One Serious Adverse Event (SAE), Medically-attended Adverse Events (MAAEs), AEs of Special Interest (AESIs) and AEs Leading to Study Withdrawal | From Day 0 up to the end of study (Day 365)
Proportion of Participants With Clinically Significant Safety Laboratory Abnormalities | At screening, and after dosing, at Days 0, 7, and 28
Proportion of Participants With RSV/A, RSV/B, hMPV/A and hMPV/B Specific NAbs RSV and hMPV IgG Prefusion F Protein-specific Antibody Titers, RSV and hMPV IgG prefusion F protein-specific antibody titers | At Days 0, 7, 180, and 365
Geometric Fold Rise (GMFR) in Serum for Anti-RSV/A, RSV/B, hMPV/A and hMPV/B Specific NAb | From Day 0 up to Day 180
  Serum samples will be collected and the titers of serum neutralization antibodies will be assessed. GMFR is defined as the geometric mean of the ratio of concentration at specified timepoints after vaccination divided by concentration at baseline (Day 0).
GMFR in Serum for RSV and hMPV IgG Prefusion F Protein-specific Antibody Titers | From Day 0 up to Day 180
  GMFR is defined as the geometric mean of the ratio of concentration at specified timepoints after vaccination divided by concentration at baseline (Day 0).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - CenExcel RCA, Hollywood, Florida
  - CenExcel ACMR, Atlanta, Georgia
  - Meridien Clinical Research, Omaha, Nebraska
  - PanAmerican Clinical Research, Brownsville, Texas

IPD SHARING:
Plan to Share IPD: No